CLINICAL TRIAL: NCT03820804
Title: Trends in Nutritional Status of Patients With Phenylketonuria
Brief Title: Nutritional Status in Phenylketonuria
Acronym: TNSPKU
Status: Completed | Type: Observational
Sponsor: Universidade do Porto (Other)
Collaborators: Centro Hospitalar do Porto (Other); BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: Nutrition_PKU
Record Dates: First submitted 2018-10-19; First posted 2019-01-29 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2018-12

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias | interventions — Diet; sapropterin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Diet-treated: Patients with Phenylketonuria under dietary treatment.
  Interventions: Other: Diet
- Sapropterin-treated: Patients with Phenylketonuria under sapropterin treatment.
  Interventions: Drug: Sapropterin

INTERVENTIONS:
Other: Diet — A specific dietary treatment for patients with Phenylketonuria.
  Other Names: Dietary treatment
  Groups: Diet-treated
Drug: Sapropterin — A pharmacological treatment for patients with Phenylketonuria, used alone or in combination with dietary treatment.
  Other Names: Tetrahydrobiopterin
  Groups: Sapropterin-treated

SUMMARY:
In the era of Phenylketonuria (PKU) newborn screening, early diagnosis in the neonatal period and prompt treatment institution has protected patients from developing severe and irreversible mental retardation. The main objective of the treatment is to prevent a chronic elevation of blood Phe concentrations, which together with reduced tyrosine concentrations may increase the risk of neurologic damage. In order to achieve this purpose, the mainstay of treatment is a special diet characterized by a natural protein restriction, supplemented with protein substitutes and special low protein foods.

The requirement to optimize growth and body composition, usually result in dietary prescriptions that are high in carbohydrate (>60% of energy intake), to promote anabolism, considering the synthetic properties of this special diet. Some studies have described a high risk of developing overweight and obesity. Although there is a tendency for a higher incidence in females, it seems that the prevalence in PKU patients follows the same trend as the general population. However, there are limited studies published so far and no longitudinal studies are available describing current practice and its impact on the prevalence of overweight and obesity; neither its consequences in terms of metabolic syndrome or cardiometabolic markers.

Recently, sapropterin dihydrochloride, which is the synthetic form of Phenylalanine Hydroxylase cofactor, is available in Portugal for patients with PKU. In practice, the sapropterin treated patients increase their natural protein intake, minimizing the synthetic characteristics of the diet. While there is a need for patient re-education about the practicalities of meeting their nutritional needs, scientific evidence about the nutritional status impact of diet liberalization is inadequate.

This study aims to test the following hypothesis:

1. Global nutritional status is not significantly affected in patients with PKU under exclusive dietary treatment.
2. There is a trend for increased rates of overweight and obesity in patients with PKU from 2009 and we consider this will continue to increase.
3. The start of sapropterin treatment allows a higher natural protein intake in patients with PKU that significantly targets nutritional status in at least one of its components (anthropometry, body composition or biochemistry).

DETAILED DESCRIPTION:
At the Centro Hospitalar do Porto (Reference Centre for the treatment of Inherited Metabolic Diseases) the annual nutritional status evaluation routinely generates data on anthropometry, body composition, blood pressure, nutritional intake and clinical biochemistry. Since 2009, all this information is recorded for all the patients with PKU under follow-up.

For the purpose of this project, data will be collected, from 2009 until 2018, using a minimum of 5 annual nutritional status evaluations per patient. The project will be able to compare the longitudinal evolution of nutritional status in exclusively diet treated patients (period between 2009 and 2014) with a subgroup of patients already under sapropterin treatment in the period between 2015 and 2018. Genotype is available for all patients with PKU under follow-up at Centro Hospitalar do Porto. However, the decision for starting sapropterin treatment was based on the results from a sapropterin-loading test protocol, approved in 2014 by the Portuguese Society of Metabolic Disorders (not published).

For every PKU patient under follow-up at Centro Hospitalar do Porto, the information about nutritional intake is recorded in a special file that contains all the diet details collected in every appointment. In that way, for the purpose of the annual nutritional status evaluation, every PKU patient is submitted to anthropometric and body composition evaluations, blood pressure assessment and blood samples collection for completing the hematological and biochemical measurements. Also in the same day, at the nutrition appointment, a dietary assessment is done, in order to allow further nutrition adjustments when needed. This approach allows us to know the precise nutritional ingestion in the period before all the measurements.

Data will be collected from patient databases or patient records. In the period between 2009 and 2014 there are no treatments or interventions to which the patients can be randomly assigned, as no specific treatment is the focus of the project. In the period between 2015 and 2018, patients will be divided in two groups based on treatment modalities: diet-treated only or sapropterin treatment. However, their assignment in each group does not have any influence of the project itself. The inclusion in one of the two groups will be decided based on the results of the sapropterin loading test done previously within the clinical routine protocol. Patients will be identified only by a number and only medical data will be collected. No directly or indirectly nominative data will be collected and data will be anonymous.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PKU.
* With all the clinical data available since 2009.
* Have completed the annual routine nutritional status evaluation in the periods 2009/2010, 2011/2012, 2013/2014, 2015/2016 and 2017/2018.
* Maintaining a follow-up at Centro Hospitalar do Porto.

Exclusion Criteria:

* Lost of follow-up.
* Not have completed at least one full evaluation in each time period: 2009/2010, 2011/2012, 2013/2014, 2015/2016 and 2017/2018.
* Any other chronic medical condition which may affect diet or nutritional status.

Min Age: 3 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Centro Hospitalar do Porto is one Portuguese Reference Centre for the treatment of inborn errors of metabolism. A cohort of patients with Phenylketonuria is under follow-up with different treatment strategies implemented. All treatment strategies are fully reimbursed by the Portuguese health system and this project aims to evaluate the longitudinal impact of different treatment options on nutritional status outcome.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Overweight and obesity prevalence | 2009-2018
  To determine the prevalence of overweight and obesity.
Overweight and obesity incidence | 2009-2018
  To determine the incidence of overweight and obesity.

SECONDARY OUTCOMES:
Metabolic syndrome prevalence | 2009-2018
  To determine the change of the prevalence of metabolic syndrome in patients.
Metabolic syndrome incidence | 2009-2018
  To determine the incidence of metabolic syndrome in patients.
Body composition using bioelectrical impedance analysis | 2009-2018
  To describe the body composition evolution (fat mass, fat-free mass and phase angle) throughout the 10 years of the study.
Metabolic control (blood phenylalanine concentration) | 2009-2018
  To describe the evolution of metabolic control in patients.
Metabolic control (blood phenylalanine concentration) and sapropterin | 2015-2018
  To describe the evolution of metabolic control (blood phenylalanine concentrations) in patients under sapropterin treatment during the period between 2015 and 2018.
Phenylalanine intake and sapropterin | 2015-2018
  To understand the impact of sapropterin treatment on phenylalanine intake (mg of phenylalanine/day) during the period between 2015 and 2018.

CONTACTS AND LOCATIONS:
Overall Officials: Júlio C Rocha, PhD, Principal Investigator — Centro Hospitalar do Porto
Locations (1):
- Centro Hospitalar Universitário do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
A detailed list of the variables to be collected can be shared with other researchers.

REFERENCES:
- [Background] MacDonald A, Rocha JC, van Rijn M, Feillet F. Nutrition in phenylketonuria. Mol Genet Metab. 2011;104 Suppl:S10-8. doi: 10.1016/j.ymgme.2011.08.023. Epub 2011 Sep 2. PMID 21944460
- [Background] Rocha JC, van Spronsen FJ, Almeida MF, Soares G, Quelhas D, Ramos E, Guimaraes JT, Borges N. Dietary treatment in phenylketonuria does not lead to increased risk of obesity or metabolic syndrome. Mol Genet Metab. 2012 Dec;107(4):659-63. doi: 10.1016/j.ymgme.2012.10.006. Epub 2012 Oct 16. PMID 23137570
- [Background] Dokoupil K, Gokmen-Ozel H, Lammardo AM, Motzfeldt K, Robert M, Rocha JC, van Rijn M, Ahring K, Belanger-Quintana A, MacDonald A. Optimising growth in phenylketonuria: current state of the clinical evidence base. Clin Nutr. 2012 Feb;31(1):16-21. doi: 10.1016/j.clnu.2011.09.001. Epub 2011 Sep 29. PMID 21959353
- [Background] Rocha JC, MacDonald A, Trefz F. Is overweight an issue in phenylketonuria? Mol Genet Metab. 2013;110 Suppl:S18-24. doi: 10.1016/j.ymgme.2013.08.012. Epub 2013 Aug 31. PMID 24055312
- [Background] MacDonald A, Ahring K, Dokoupil K, Gokmen-Ozel H, Lammardo AM, Motzfeldt K, Robert M, Rocha JC, van Rijn M, Belanger-Quintana A. Adjusting diet with sapropterin in phenylketonuria: what factors should be considered? Br J Nutr. 2011 Jul;106(2):175-82. doi: 10.1017/S0007114511000298. PMID 21466737
- [Background] Rocha JC, van Spronsen FJ, Almeida MF, Ramos E, Guimaraes JT, Borges N. Early dietary treated patients with phenylketonuria can achieve normal growth and body composition. Mol Genet Metab. 2013;110 Suppl:S40-3. doi: 10.1016/j.ymgme.2013.10.009. Epub 2013 Oct 22. PMID 24183791
- [Background] Gokmen Ozel H, Ahring K, Belanger-Quintana A, Dokoupil K, Lammardo AM, Robert M, Rocha JC, Almeida MF, van Rijn M, MacDonald A. Overweight and obesity in PKU: The results from 8 centres in Europe and Turkey. Mol Genet Metab Rep. 2014 Nov 16;1:483-486. doi: 10.1016/j.ymgmr.2014.11.003. eCollection 2014. PMID 27896128
- [Background] Rocha JC, van Rijn M, van Dam E, Ahring K, Belanger-Quintana A, Dokoupil K, Gokmen Ozel H, Lammardo AM, Robert M, Heidenborg C, MacDonald A. Weight Management in Phenylketonuria: What Should Be Monitored. Ann Nutr Metab. 2016;68(1):60-5. doi: 10.1159/000442304. Epub 2015 Nov 25. PMID 26598928